CLINICAL TRIAL: NCT03013283
Title: Descriptional Study of the Side Effects Related to the Use of the Interface in Home Care Patients Treated for at Least 3 Months by Continuous Positive Pressure or Non-Invasive Ventilation.
Brief Title: CPAP and NIV Interfaces : Side-effects in Home Care Patients
Acronym: InterfaceVent
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL16_0337
Record Dates: First submitted 2016-12-23; First posted 2017-01-06 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2019-04

CONDITIONS: Interface, Mask; Continuous Positive Airway Pressure (CPAP); Non Invasive Ventilation (NIV); Hyperventilation Anxiety; Sleep Apnea Syndrome (OSAS)
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: self questionnaire — * Interface side effects and degree of satisfaction of the patients
  * Technician evaluation and device measures.

SUMMARY:
Home ventilation techniques consist mainly of two techniques, Continuous Positive Airway Pressure or CPAP and Non Invasive Ventilation or NIV. Whether for CPAP or NIV, pressures are delivered to the patient via an interface.

The efficacy of CPAP and NIV is conditioned in part by the observance of the patients to the device. Because the comfort and degree of satisfaction of the patients to its interface is a key factor of the observance, side-effects and satisfaction of patients need to be continuously evaluated with available interfaces for CPAP and NIV treated patients.

The purpose of the research is the evaluation of interface side-effects and the degree of satisfaction of home care patients treated for at least three months with CPAP or NIV.

DETAILED DESCRIPTION:
Home ventilation techniques consist mainly of two techniques, Continuous Positive Airway Pressure or CPAP (the level of pressure delivered being constant) and Non Invasive Ventilation or NIV (pressure level varies from an expiratory pressure to an inspiratory pressure). Whether for CPAP or NIV, pressures are delivered to the patient via an interface. Many manufacturers produce interfaces and these interfaces are the subject of regular technological innovations with the introduction on the market of new product ranges.

Because of the lack of dedicated and actualized studies, there is poor evidence based of difference between old and new interfaces, there is also poor evidence based of differences between manufacturer products.

The efficacy of CPAP and NIV is conditioned in part by the observance of the patients to the device. Because the comfort and degree of satisfaction of the patients to its interface is a key factor of the observance, side-effects and satisfaction of patients need to be continuously evaluated with available interfaces for CPAP and NIV treated patients.

The purpose of the research is the evaluation of interface side-effects and the degree of satisfaction of home care patients treated for at least three months with CPAP or NIV. A visual analog scale is used to assess the patient perception of its interface. A measure of the quality of life and a home care technician evaluation are performed simultaneously. Using the device manufacturer software, a measure of the observance, level of pressure and leak is realised.

A first intermediate analysis will be made after approximately 1000 inclusions (the Sleepileaks (determinants of residual excessive sleapiness), Threshleaks (high leak levels and machine adherence as defined by the American Thoracic Society) and Complileaks studies (all leaks and machine adherence as continuous variables)). A second validating analysis will be made at the end of inclusions.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age more than 18 years (inclusive)
* Patient treated with CPAP or NIV for at least three months,and eligible for care and for the reimbursement by the French Social Security rules.
* Patient presents during a scheduled home visit of the technician for the continuation of CPAP or NIV treatment according to the French Social Security rules.

Exclusion Criteria:

* Pregnancy, intention of being pregnant, breastfeeding.
* Inability to understand the nature and aims of the study or to communicate with the investigator
* Simultaneous participation in another trial with an exclusion clause to participate to an other trial.
* No affiliation to the French social security
* Loss of personal capacity resulting in state protection
* Deprivation of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included in the study corresponded to the annual cohort of patients cared by the APARD home care provider. Patients are were treated with CPAP or VIN for more than 3 months according to the criteria of care and reimbursement of the French Social Security rules.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Interface side effects and degree of satisfaction of the patients | 1 day
  During a scheduled home visit of the technician. The primary endpoint is a composite criterion corresponding to the patients' responses to a self-administered questionnaire.

SECONDARY OUTCOMES:
Identification by the technician of the problems of pain | 1 day
  During a scheduled home visit of the technician : Identification by the technician of the problems of pain, erythema and leak, localization of these problems.
Percentage of patients with oxygen therapy, heated humidifier, chinstrap. | 1 day
  During a scheduled home visit of the technician : Percentage of patients with oxygen therapy, heated humidifier, chinstrap.
Collection by technician of the type of interface | 1 day
  During a scheduled home visit of the technician : Collection by technician of the type of interface (nasal pillows, nasal and oronasal, custom made interface), manufacturer name and interface size, type (CPAP/NIV) and manufacturer name of the device.
Compliance | 1 day
  During a scheduled home visit of the technician : Device software data: compliance (hour per day) over the last 3 months
Average level of intentional or unintentional leakage | 1 day
  During a scheduled home visit of the technician : Device software data: average level of intentional or unintentional leakage (l/min)
Residual AHI | 1 day
  During a scheduled home visit of the technician : Device software data: residual AHI (event/hour)
Average pressure level and pressure | 1 day
  During a scheduled home visit of the technician :Device software data: average pressure level and pressure at the 90/95th percentile (cmH2O).
Patient quality of life questionnaire | 1 day
  Patient quality of life questionnaire (EQ-5D 3L, Epworth).
Date of first installation of the first ventilation device | 1 day
  Date of first installation of the first ventilation device
Proportion of patient responding to self-help questionnaire without assistance | 1 day
  Proportion of patient responding to self-help questionnaire without assistance
Proportion of patients able to position the interface without assistance | 1 day
  Proportion of patients able to position the interface without assistance
Time taken by the patient and the technician to answer the patient's self-questionnaire and the technician record respectively. | 1 day
  Time taken by the patient and the technician to answer the patient's self-questionnaire and the technician record respectively.
Proportion of patient waiting for a new interface | 1 day
  Proportion of patient waiting for a new interface
Proportion of patients wishing to participate in research on the subject. | 1 day
  Proportion of patients wishing to participate in research on the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Dany JAFFUEL, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - CHU Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rotty MC, Mallet JP, Suehs CM, Martinez C, Borel JC, Rabec C, Bourdin A, Molinari N, Jaffuel D. Is the 2013 American Thoracic Society CPAP-tracking system algorithm useful for managing non-adherence in long-term CPAP-treated patients? Respir Res. 2019 Sep 12;20(1):209. doi: 10.1186/s12931-019-1150-7. PMID 31514751
- [Result] Rotty MC, Suehs CM, Mallet JP, Martinez C, Borel JC, Rabec C, Bertelli F, Bourdin A, Molinari N, Jaffuel D. Mask side-effects in long-term CPAP-patients impact adherence and sleepiness: the InterfaceVent real-life study. Respir Res. 2021 Jan 15;22(1):17. doi: 10.1186/s12931-021-01618-x. PMID 33451313
- [Derived] Vidal C, Mallet JP, Skinner S, Gilson R, Gaubert O, Prigent A, Gagnadoux F, Borel JC, Bourdin A, Molinari N, Jaffuel D. Positive Airway Pressure-Related Aerophagia in Obstructive Sleep Apnea: Results from the InterfaceVent Real-Life Study. J Clin Med. 2025 Sep 11;14(18):6424. doi: 10.3390/jcm14186424. PMID 41010628
- [Derived] Vidal C, Bertelli F, Mallet JP, Gilson R, Borel JC, Gagnadoux F, Skinner S, Bourdin A, Molinari N, Jaffuel D. Added value of technician intervention to improve mask management for apneic patients treated with long-term CPAP. Sleep Breath. 2025 Feb 28;29(1):117. doi: 10.1007/s11325-025-03279-2. PMID 40019603
- [Derived] Vidal C, Bertelli F, Mallet JP, Gilson R, Borel JC, Gagnadoux F, Bourdin A, Molinari N, Jaffuel D. Mask side-effects are related to gender in long-term CPAP: results from the InterfaceVent real-life study. Respir Res. 2024 Sep 6;25(1):331. doi: 10.1186/s12931-024-02965-1. PMID 39243031
- See also: InterfaceVent on the Open Science Framework — https://osf.io/sy3nq/